CLINICAL TRIAL: NCT06492395
Title: A Multicentre, Randomised Controlled Study of Lenvatinib Plus Drug-eluting Bead Transarterial Chemoembolization and Hepatic Arterial Infusion Chemotherapy With FOLFOX Regimen Versus Lenvatinib Plus Drug-eluting Bead Transarterial Chemoembolization for Hepatocellular Carcinoma Larger Than 7 cm With Portal Vein Tumor Thrombosis
Brief Title: Lenvatinib Plus DEB-TACE and HAIC vs. Lenvatinib Plus DEB-TACE for Large HCC With PVTT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-18
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: hepatocellular carcinoma; lenvatinib; transarterial chemoembolization; drug-eluting bead; hepatic arterial infusion chemotherapy; portal vein tumor thrombosis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Len+DEB-TACE+HAIC (Experimental): Patients will receive the combination treatment of Len+DEB-TACE+HAIC.
  Interventions: Combination Product: Len+DEB-TACE+HAIC
- Len+DEB-TACE (Active Comparator): Patients will receive the combination treatment of Len+DEB-TACE.
  Interventions: Combination Product: Len+DEB-TACE

INTERVENTIONS:
Combination Product: Len+DEB-TACE+HAIC — For DEB-TACE, superselective catheterization is performed and DEBs loaded with pirarubicin is use for chemoembolization. The embolization end point was blood stasis of the tumor-feeding arteries. In order to reduce the risk of complications, the embolization end point was not achieved in the initial TACE but in the second or third TACE session.
  After each chemoembolization, the microcatheter is reserved at the main hepatic tumor-feeding artery. The FOLFOX-based regimen is intra-arterially administered.
  During follow-up, the treatment of DEB-TACE and/or HAIC will be repeated for viable tumors based on the evaluation of the follow-up laboratory and imaging examination.
  Lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. qd will be started with 7 days after the first DEB-TACE+HAIC.
  Arms: Len+DEB-TACE+HAIC
Combination Product: Len+DEB-TACE — For DEB-TACE, superselective catheterization is performed and DEBs loaded with pirarubicin is use for chemoembolization. The embolization end point was blood stasis of the tumor-feeding arteries. In order to reduce the risk of complications, the embolization end point was not achieved in the initial TACE but in the second or third TACE session. During follow-up, the treatment of DEB-TACE will be repeated for viable tumors based on the evaluation of the follow-up laboratory and imaging examination.
  Lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. qd will be started with 7 days after the first DEB-TACE+HAIC.
  Arms: Len+DEB-TACE

SUMMARY:
This study is conducted to evaluate the efficacy and safety of lenvatinib plus transarterial chemoembolization (TACE) with drug-eluting beads (DEB-TACE) and hepatic artery infusion chemotherapy (HAIC) with FOLFOX regemen (Len+DEB-TACE+HAIC) versus lenvatinib plus DEB-TACE (Len+DEB-TACE) for large hepatocellular carcinoma (> 7cm) with portal vein tumor thrombosis (PVTT).

DETAILED DESCRIPTION:
This is a multicenter, prospective and randomized study to evaluate the efficacy and safety of Len+DEB-TACE+HAIC compared with Len+DEB-TACE for unresectable large HCC (>7cm) with PVTT.

178 patients with large HCC (> 7cm) and PVTT will be enrolled in this study. The patients will receive either Len+DEB-TACE+HAIC or Len+DEB-TACE using an 1:1 randomization scheme. In the Len+DEB-TACE+HAIC arm, the microcatheter will be reserved at the main hepatic tumor-feeding artery after DEB-TACE and chemotherapy drugs (oxaliplatin, fluorouracil and leucovorin; FOLFOX-based regimen) will be intra-arterially administered though the microcatheter. DEB-TACE+HAIC treatments can be repeated based on the evaluation of follow-up laboratory and imaging examination by the multidisciplinary team. In the Len+DEB-TACE arm, patients will be treated with DEB-TACE alone. TACE treatment can be repeated based on the evaluation of follow-up laboratory and imaging examination by the multidisciplinary team. In both arms, lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. qd will be started within 7 days after the first DEB-TACE+HAIC/DEB-TACE.

The primary end point of this study is time to progression (TTP). The secondary endpoints are tumor response (objective response rate and disease control rate), overall survival (OS), and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of HCC
* the largest intrahepatic lesion >7 cm
* presence of PVTT on imaging
* tumor recurrence after curative treatment (hepatectomy or ablation) is eligible for enrollment
* Eastern Cooperative Oncology Group performance status ≤1
* Child-Pugh class A/B
* adequate hematologic and organ function, with leukocyte count>3.0×10^9/L, neutrophil count>1.5×10^9/L, platelet count≥75×10^9/L, hemoglobin 85 g/L, alanine transaminase and aspartate transaminase≤5×upper limit of the normal, creatinine clearance rate≤1.5×upper limit of the normal
* life expectancy of at least 3 months

Exclusion Criteria:

* Diffuse HCC
* accompanied with vena cava tumor thrombus
* central nervous system involvement
* previous treatment with TACE, HAIC, TAE, radiotherapy, or systemic therapy
* organ (heart and kidneys) dysfunction, unable to tolerate TACE or HAIC treatment
* history of other malignancies
* uncontrollable infection
* history of HIV
* history of organ or cells transplantation
* prothrombin time prolongation >4 s

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to progression (TTP) | 2 years
  The time from date of randomization until the first occurrence of disease progression (according to mRECIST).

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  The proportion of patients with the best response of complete response (CR) or partial response (PR) according to mRECIST.
Disease control rate (DCR) | 2 years
  The proportion of patients with the best response of CR, PR, or stable disease (SD) according to mRECIST.
Overall survival (OS) | 3 years
  The time from date of randomization to death due to any cause.
Adverse Events (AEs) | 3 years.
  Number of patients with AEs assessed by Common Terminology Criteria for Adverse Events v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided